CLINICAL TRIAL: NCT04841369
Title: A Randomized,Blind, Positive-controlled Phase III Clinical Trial to Evaluate the Safety and Immunogencity of 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT） in Healthy People Aged 6 Weeks and Above
Brief Title: Phase III Clinical Trial of a Candidate PCV13 in Healthy People Aged 6 Weeks and Above (PICTPCV13i)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS-CTP-PCV-III
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2022-10

CONDITIONS: Pneumococcal Infections; Streptococcal Infections; Bacterial Infections
Keywords: PCV13; 13 valent Pneumococcal conjugate vaccine; Pneumococcal Infections; Safety; Immunogenicity
MeSH Terms: conditions — Pneumococcal Infections; Streptococcal Infections; Bacterial Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 1A (Experimental): Subjects received four doses of PCV13i at 2 months of age (At least 6 weeks old)
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- 1B (Active Comparator): Subjects received four doses of PCV13 at 2 months of age (At least 6 weeks old)
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 2A (Experimental): Subjects received four doses of PCV13i at 3 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- 3A (Experimental): Subject received three doses of PCV13i at 7 to 11 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- 3B (Active Comparator): Subject received three doses of PCV13 at 7 to 11 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 4A (Experimental): Subjects received two doses of PCV13i at 12 to 23 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- 4B (Active Comparator): Subjects received two doses of PCV13 at 12 to 23 months of age
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine
- 5A (Active Comparator): Subjects received one dose of PCV13i at 2 to 5 years old.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT）
- 5B (Active Comparator): Subjects received one dose of PCV13 at 2 to 5 years old.
  Interventions: Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine

INTERVENTIONS:
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine（CRM197,TT） — 0.5mL,Intramuscular
  Other Names: PCV13i
  Arms: 1A; 2A; 3A; 4A; 5A
Biological: 13-Valent Pneumococcal Polysaccharide Conjugate Vaccine — 0.5mL,Intramuscular
  Other Names: Prevnar
  Arms: 1B; 3B; 4B; 5B

SUMMARY:
Streptococcus pneumoniae is a major cause of morbidity and mortality in children worldwide, resulting in up to 1 million pediatric deaths every year.Since the licensure of PCV7 and PCV13,the reported overall decline in invasive pneumococcal disease in hospitalized children younger than 5 years several years is approximately 60% in Western countries.This is a single center,blind, randomized, positive-controlled clinical trial.The purpose of this study is to preliminary evaluate the safety of PCV13i vaccine in subjects at age of 7 months and above,and to investigate the safety and immunogenicity of PCV13i vaccine at age of 2 and 3 months,compared to PCV13.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of 2 months (minimum 6 weeks), 3 months , 7 months and above;
* Willing to provide proof of identity;
* Without vaccination history of pneumococcal vaccine;
* None-pregnancy or do not plan to pregnancy recently;;
* Volunteers of 18 years old and above who have the ability to understand clinical studie progress and sign informed consent;
* Volunteers of 8-17 years old and their guardians who willing sign informed consent;
* Able to understand and sign the informed consent by their guardians or trustees for the volunteers of 8 years old and below;
* Able and willing comply with the requirements of the protocol

Exclusion Criteria:

* Volunteers whose axillary body temperature was >37.0# before vaccination
* Volunteers who suffered from Congenital malformation or developmental disorder, genetic defect, severe malnutrition, etc;
* Volunteers who has a history of epilepsy, convulsions or psychosis;
* Allergic person;
* Any prior administration of blood products in last 3 month;
* Any prior administration of other research medicines in last 1 month;
* Plans to participate in or is participating in any other drug clinical study;
* Any prior administration of attenuated live vaccine in last 14 days;
* Any prior administration of subunit or inactivated vaccines in last 7 days;
* Had fever before vaccination, Volunteers with temperature >37.0°C on axillary setting;
* According to the investigator's judgement, the subjects have any other factors that make them unfit to enroll the clinical trial

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3420 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Safety of PCV13i in preventing pneumococcal infections | Within 7 days post each vaccination
  Occurance of adverse reactions in all subjects
Safety of PCV13i in preventing pneumococcal infections | Within 30 days post each vaccination
  Occurance of adverse reactions in all subjects
Immunogenicity of PCV13i in subjects of 2 months (at least 6 weeks) old (Arm 1A-1B) | 30 days post three doses
  Serotype-specific seropositivity rates of Immunoglobulin G GMC concentrations above 0.35ug/ml
Immunogenicity of PCV13i in subjects of 7 to 11 months old (Arm 4A-4B) | 30 days post three doses
  Serotype-specific seropositivity rates of Immunoglobulin G GMC concentrations above 0.35ug/ml
Immunogenicity of PCV13i in subjects of 12 months to 5 years old (Arm 5A, 5B, 6A, 6B) | 30 days post last dose of vaccination
  Serotype-specific seropositivity rates of Immunoglobulin G GMC concentrations above 0.35ug/ml
Immunogenicity of PCV13i in subjects of age 50 years old and above (Arm 6A, 6B, 7A, 7B) | 30 days post vaccination
  Serotype-specific seropositivity rates of Immunoglobulin G GMC concentrations above 0.35ug/ml

SECONDARY OUTCOMES:
Immuogenicity in terms of GMT in subjects of 2 months (at least 6 weeks) old (Arm 1A-1B) | 30 days post three doses
  GMT of serotype-specific OPA antibody with the titer of ≥1:8 ratio
Immunogenicity in terms of IgG concentration in subjects of 2 months (at least 6 weeks) old (Arm 1A-1B) | 30 days post three doses
  Serotype-specific Immunoglobulin G with a concentration of ≥1.0μg/ml
Safety of PCV13i in terms of in subjects of 2 months (at least 6 weeks) old (Arm 1A-1B) | 6 months post one to three doses of vaccination
  Occurance of SAE in subjects of this age group
Immuogenicity in terms of GMT in subjects of 7 to 11 months old (Arm 3A-3B) | 30 days post two doses
  GMT of serotype-specific OPA antibody with the titer of ≥1:8 ratio
Immuogenicity in terms of GMT in subjects of 12 months to 5 years old (Arm 4A, 4B, 5A, 5B) | 30 days post last dose of vaccination
  GMT of serotype-specific OPA antibody with the titer of ≥1:8 ratio
Immunogenicity in terms of IgG concentration in subjects of 7 to 11 months old (Arm 3A-3B) | 30 days post two doses
  Serotype-specific Immunoglobulin G with a concentration of ≥1.0μg/ml
Immunogenicity in terms of IgG concentration in subjects of 12 months to 5 years old (Arm 4A, 4B, 5A, 5B) | 30 days post last dose of vaccination
  Serotype-specific Immunoglobulin G with a concentration of ≥1.0μg/ml
Safety of PCV13i in terms of SAE in subjects of 7 to 11 months old (Arm 3A-3B) | 6 months post two doses
  Occurance of SAE in subjects of this age group
Safety of PCV13i in terms of SAE in subjects of 12 months to 5 years old (Arm 4A, 4B, 5A, 5B) | 6 months post last dose of vaccination
  Occurance of SAE in subjects of this age group

CONTACTS AND LOCATIONS:
Overall Officials: Shengli Xia, Principal Investigator — Henan Province Center for Disease Control and Prevention
Locations (1):
- Neihuang Center for Disease Control and Prevention, Anyang, Henan, China